CLINICAL TRIAL: NCT05907330
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase 2 Study to Evaluate the Efficacy and Safety of CU104 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Phase 2 Study of CU104 in Moderate-Severe Ulcerative Colitis
Acronym: UC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Curacle Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CU104-P2-01
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CU104 (Experimental): CU104 100 mg three capsules a day .
  Interventions: Drug: CU104
- Placebo (Placebo Comparator): Placebo three capsules a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CU104 — CU104 will administer the study drug once a day after a meal
  Arms: CU104
Drug: Placebo — Placebo will administer the study drug once a day after a meal
  Arms: Placebo

SUMMARY:
The study is designed to investigate efficacy and safety of CU104 in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 to 80 years.
4. Males and female patients with clinical diagnosis of ulcerative colitis ≥3 months prior to Screening.
5. Active, moderate to severe ulcerative colitis, as defined by the modified Mayo score of 5 to 9, including an endoscopy sub-score of at least 2.
6. For females of reproductive potential: Use of highly effective contraception for at least 1 month prior to Screening and agreement to use such method during study participation and for an additional 8 weeks after the last dose.
7. For males of reproductive potential: Use of condoms or other methods to ensure effective contraception during study participation and for an additional 8 weeks after the last dose.

Exclusion Criteria:

1. Received any of the following, prior to randomization for the treatment of UC:

   * Corticosteroids (intravenous or rectal administration) or 5-aminosalicylic acid (rectal administration) within 3 weeks;
   * Janus kinase (JAK) inhibitors within 2 weeks;
   * Cyclosporine, mycophenolate, tacrolimus, methotrexate, azathioprine, or 6- mercaptopurine within 4 weeks;
   * Anti-TNF-α biologics within 8 weeks; or
   * Any other commercially approved biologic agent or targeted small molecule within 8 weeks or within 5 half-lives whichever is longer.
2. Have been diagnosed with UC limited to the rectum (disease which extends < 15 cm above the anal verge).
3. Received orally administered 5-aminosalicylic acid (ASA), sulfasalazine, or low-dose corticosteroids (prednisolone ≤20 mg/day or its equivalent) on a stable regimen (i.e., no changes in drug or dose) for <4 weeks prior to randomization. The doses must remain stable until the end of study treatment (with possible exception for tapering steroid dose after 8 weeks).
4. Received any other concomitant medications for UC on a stable regimen (i.e., no changes in drug or dose) for <2 weeks or 5 half-lives, whichever is longer.
5. Presence of Crohn's disease, indeterminate colitis, ischemic colitis, fulminant colitis, ulcerative proctitis, or toxic megacolon.
6. Previous extensive colonic resection (subtotal or total colectomy).
7. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
8. Evidence of or treatment for, Clostridium difficile infection or other pathogenic bowel infection within 60 days or for another intestinal pathogen within 30 days prior to randomization.
9. Active viral infection with HIV, Hepatitis B, or Hepatitis C.
10. Clinically significant, active extraintestinal infection (e.g., pneumonia, pyelonephritis).
11. History of cancer, including solid tumors and hematological malignancies (except basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved).
12. History of any clinically significant medical condition that, in the investigator's opinion, would preclude participation in the study (e.g., End-stage renal disease (ESRD), severe liver diseases).
13. Has unstable angina, myocardial infarction, transient ischemic attack, cerebral infarction, coronary artery bypass surgery, or transluminal coronary angioplasty within 6 months before screening.
14. Other clinically significant abnormal lab values per Investigator's judgement.
15. Pregnancy or lactation.
16. Treatment with another investigational drug or other intervention within 30 days prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with clinical remission at Week 8 | Week 8
  Clinical remission is defined as a modified Mayo score o to 2

IPD SHARING:
Plan to Share IPD: No